CLINICAL TRIAL: NCT01757431
Title: The Safety and Efficacy of Eculizumab in Japanese Patients With Atypical Hemolytic Uremic Syndrome (aHUS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C11-005J
Record Dates: First submitted 2012-12-04; First posted 2012-12-31 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Atypical Hemolytic Uremic Syndrome (aHUS)
MeSH Terms: conditions — Atypical Hemolytic Uremic Syndrome | interventions — eculizumab

ARMS (1):
- ECULIZUMAB (Other)
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab

SUMMARY:
Protocol is intended to characterize the overall safety and tolerability of eculizumab in this population.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with diagnosis of aHUS who have been receiving eculizumab by personal importation (specific eligibility criteria below do not apply) Or,
2. Patients with current clinical manifestations of aHUS who meet the following criteria:

   1. Patient with diagnosis of aHUS with or without an identified complement regulatory protein genetic abnormality or anti-complement factor antibody and for whom other known etiologies of hemolytic uremic syndrome (HUS) have been ruled out as confirmed in the Exclusion Criteria
   2. Patient (and legal guardian if patient is not an adult) willing and able to give written informed consent and assent (or verbal assent if patient is unable to read or write)
   3. Patient at least 1 month of age and body weight ≥5 kg
   4. Platelet count at screening < lower limit of normal (LLN)
   5. Signs or symptoms of hemolysis (i.e., lactate dehydrogenase (LDH) ≥ 1.5x upper limit of normal (ULN) and Hemoglobin ≤ LLN) at start of current aHUS event
   6. Serum Creatinine (SrCr) level ≥ ULN at screening (patient requiring dialysis for acute renal failure also eligible)
   7. Female patient of childbearing potential practicing an effective, reliable and medically approved contraceptive regimen during the entire duration of the study, including the Follow-up Period. At the time of the last follow-up visit, patient must agree to continue to use adequate contraception methods for up to 5 months following discontinuation of eculizumab treatment
   8. Able and willing to comply with study procedures

Exclusion Criteria:

Shiga-toxin producing E. coli-HUS (STEC-HUS; shiga-toxin and/or STEC positive) History of malignancy within 5 years of screening Known human immunodeficiency virus (HIV) infection Identified drug exposure-related HUS Infection-related HUS HUS related to bone marrow transplant (BMT) HUS related to vitamin B12 deficiency Known Systemic Lupus Erythematosus (SLE) or antiphospholipid antibody positivity or syndrome Chronic dialysis (defined as dialysis on a regular basis as renal replacement therapy for end-stage renal disease (ESRD)) Patients with a confirmed diagnosis of sepsis defined as positive blood cultures within 7 days of the screening visit and not treated with antibiotics to which the organism is sensitive Presence or suspicion of active and untreated systemic bacterial infection that, in the opinion of the Investigator confounds an accurate diagnosis of aHUS or impedes the ability to manage the aHUS disease Pregnancy or lactation Unresolved systemic meningococcal disease Any medical or psychological condition that, in the opinion of the investigator, could increase patient's risk by participating in the study or confound the outcome of the study Patients receiving chronic intravenous immunoglobulin (IVIG) within 8 weeks unless for unrelated medical condition (e.g., hypogammaglobulinemia) or chronic rituximab therapy within 12 weeks of the screening visit Patients receiving other immunosuppressive therapies such as steroids, calcineurin inhibitors (mTOR), (e.g., cyclosporine or tacrolimus) are excluded unless: [1] part of an established post-transplant anti-rejection regimen, or [2] patient has confirmed anti-Complement Factor Antibodies requiring immunosuppressive therapy or [3] steroids are used for a condition other than aHUS (e.g., asthma) Prior eculizumab use, hypersensitivity to eculizumab, to murine proteins or to one of the excipients Inclusion in any other investigational intervention trial except this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-05-16 (Actual); Primary Completion 2013-09-24 (Actual); Study Completion 2013-09-25 (Actual)

PRIMARY OUTCOMES:
Adverse events and serious adverse events and their severity and relationship to the drug | 12 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Nagano Red Cross Hospital, Nagano
  - Tokyo Medical and Dental University Hospital, Tokyo

REFERENCES:
- [Derived] Pugh D, O'Sullivan ED, Duthie FA, Masson P, Kavanagh D. Interventions for atypical haemolytic uraemic syndrome. Cochrane Database Syst Rev. 2021 Mar 23;3(3):CD012862. doi: 10.1002/14651858.CD012862.pub2. PMID 33783815